CLINICAL TRIAL: NCT01377129
Title: Reconstruction of the Anterior Cruciate Ligament: a Comparative MRI Study Evaluating Residual Rotational Laxity for Single Versus Double Bundle Surgical Techniques
Brief Title: Anterior Cruciate Ligament Reconstruction: Residual Rotational Laxity for Single Versus Double Bundle Techniques
Acronym: LCA IRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrolment proved to be more difficult than foreseen and was stopped at 46 inclusions.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2011/PM-03; 2011-A00465-36 (Other: RCB number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Residual Rotational Laxity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Bundle (Active Comparator): These patients are operated using a single bundle technique.
  Interventions: Procedure: Single bundle anterior cruciate ligament reconstruction
- Double bundle (Experimental): These patients are operated using a double bundle technique.
  Interventions: Procedure: Double bundle anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: Single bundle anterior cruciate ligament reconstruction — Single bundle anterior cruciate ligamentoplasty
  Arms: Single Bundle
Procedure: Double bundle anterior cruciate ligament reconstruction — Double bundle anterior cruciate ligamentoplasty
  Arms: Double bundle

SUMMARY:
The main objective of this study is to compare, using MRI measures with a specialized splint, the persistent rotatory laxity after anterior cruciate ligament reconstruction using single bundle and double bundle surgical techniques, between the seventh and eighth months after surgery, and for different degrees of knee flexion (0 °, 20 °, 40 °, 60 °).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 24 months of follow-up
* The patient requires reconstruction of the anterior cruciate ligament due to rupture confirmed by MRI

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient require a single bundle, "KJ-type" surgical technique
* Contra-indication for MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Residual rotational laxity during MRI | 7-8 months post-op
  Residual rotational laxity is defined as the difference between the operated knee and the non-operated knee for "D", where D is the distance between the posterior tibial cortex and the center of the circle which forms the lateral femoral condyle. D will be evaluated at 4 angles of flexion (0°, 20°, 40° and 60°) and evaluated as a repeated measure.

SECONDARY OUTCOMES:
Lysholm score | 7-8 months
International Knee Documentation Committee score | 7-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Marchand, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France